CLINICAL TRIAL: NCT05078008
Title: The Role of Balneotherapy in Older Adults With Chronic Low Back Pain: a Biopsychosocial Approach at São Pedro do Sul Thermal Baths
Brief Title: The Role of Balneotherapy in Older Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Termalistur - Termas de Sao Pedro do Sul, E.M., S.A. (Other)
Collaborators: Universidade do Porto (Other); Aveiro University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Termalistur
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low Back Pain; Older Adults; Health Resort Medicine; Quality of Life
Keywords: Balneotherapy; Chronic Low Back Pain; Older adults; Health Resort Medicine; Quality of Life; Thermography; Crenotherapy; Balneology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Physiotherapy modalities (Placebo Comparator)
  Interventions: Procedure: Physiotherapy modalities
- Group 2 - Physiotherapy modalities + Balneotherapy modalities (Experimental)
  Interventions: Procedure: Physiotherapy modalities; Procedure: Balneotherapy modalities

INTERVENTIONS:
Procedure: Physiotherapy modalities — parafango in the lumbar region 20min/day; High frequency Transcutaneous Electrical Nerve Stimulation (TENS), 100 Hz, 0,04-0,2mseg, 20 min/day; lumbar flexibility self-exercise plan
Procedure: Balneotherapy modalities — Immersion in a thermal pool with 15 minutes of automatic hydromassage and 15 minutes of spine flexibility exercises; thermal steam treatment to spinal column; hydromassage bath with Vichy thermal water
  Arms: Group 2 - Physiotherapy modalities + Balneotherapy modalities

SUMMARY:
The effectiveness of balneotherapy in relieving chronic low back pain has been scientifically proven. This project aims to study in what extent a Balneotherapy program in São Pedro do Sul Thermal Baths influences chronic low back pain of individuals aged 65 and above, and in what order of magnitude it happens, on which domains (functional, psychological, biophysical and socioeconomic) and it's repercussions. For that, the investigators intended to carry out a project subdivided into two tasks. The first, and the most complex, with a holistic approach, will be carried out by a randomized controlled study (RCT) with focus on the various biopsychosocial domains of patients with chronic lumbar pain. Concerning the second task, another RCT will be carried out aiming for statistically significant changes in the lumbar thermographic maps before and after treatment, as well as the theoretical framework of all the findings.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 and over
* Low back pain with or without irradiation to the lower limbs with more than 3 months of evolution
* Imaging exam of the lumbar spine that excludes neoplastic pathology or severe structural misalignments
* Availability to carry out a 14-day treatment plan

Exclusion Criteria:

* Can't read and write
* History of fracture, surgery, infection or neoplasm in the spine
* Scoliosis with a cobb angle >20
* Lower limb muscle strength or vesico-sphincter changes
* Fever, history of recent violent trauma, unexplained weight loss, night sweats, or persistent night pain
* Others: unstable angina pectoris, poorly controlled hypertension, cardiac decompensation, respiratory failure, endocrine disorder, acute febrile condition, skin infections, fecal or urinary incontinence and psychosis or decompensated neurosis

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | two weeks
  Pain assessment; From "0" (minimum - better) to "10" (maximum - worse)
Oswestry Disability Index, version 2.0 | two weeks
  Functional assessment; From "0%" (minimum - better) to "100%" (maximum - worse)
The Short Form-36 | two weeks
  Quality of life assessment; From "0" (minimum - worse) to "100" (maximum - better)
Center for Epidemiologic Studies Depression Scale | two weeks
  Depression assessment; From "0" (minimum - better) to "60" (maximum - worse)
Satisfaction with life scale - 5 items version | two weeks
  Satisfaction with life scale assessment; From "5" (minimum - worse) to "35" (maximum - better)
International Physical Activity Questionnaire - short version | two weeks
  Physical activity assessment; low values (worse) vs high values (better)
Fatigue Assessment Scale | two weeks
  Fatigue assessment; From "10" (minimum - better) to "50" (maximum - worse)
Dolorimeter | two weeks
  Pain assessment; low values (worse) vs high values (better)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson F Albuquerque, Principal Investigator — Medical Doctor
Locations (1):
- Termalistur - Termas de São Pedro do Sul, São Pedro do Sul, Viseu District, Portugal

IPD SHARING:
Plan to Share IPD: No